CLINICAL TRIAL: NCT05725434
Title: A Single-arm, Open-label, Multiple-dose, Phase 3 Study to Evaluate Usability of Subcutaneous Auto-injector of CT-P47 in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Evaluate Usability of Subcutaneous Auto-injector of CT-P47 in Patients With Active Rheumatoid Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P47 3.2
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-P47 SC (tocilizumab) (Experimental): CT-P47 (tocilizumab) by subcutaneous (SC) injection
  Interventions: Biological: CT-P47 AI (tocilizumab); Biological: CT-P47 PFS (tocilizumab)

INTERVENTIONS:
Biological: CT-P47 AI (tocilizumab) — CT-P47 (162 mg/0.9 mL) by subcutaneous (SC) injection via autoinjector (AI) at Week 0 and Week 2
Biological: CT-P47 PFS (tocilizumab) — CT-P47 (162 mg/0.9 mL) by SC injection via pre-filled syringe from Week 4 every other week or weekly (based on the clinical response by investigator's discretion) up to Week 10

SUMMARY:
This is a phase 3 study to evaluate the usability of the CT-P47 auto-injector in patients with moderate to severe active rheumatoid arthritis.

DETAILED DESCRIPTION:
CT-P47, containing the active ingredient tocilizumab, is a recombinant humanized monoclonal antibody that is being developed as a similar biological medicinal product to RoActemra/Actemra. The purpose of this study is to evaluate the usability of the CT-P47 auto-injector in patients with moderate to severe rheumatoid arthritis when co-administered with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female aged 18 to 70 years old, both inclusive.
* Patient must be able and willing to self-administer SC injections.
* Patient has had a diagnosis of RA according to the 2010 ACR/EULAR classification criteria (Aletaha et al., 2010) for at least 24 weeks prior to the first administration of the study drug (Day 1).

Exclusion Criteria:

* Patient who has previously received investigational or licensed product; targeted synthetic DMARD(s) (e.g., tofacitinib, baricitinib) for the treatment of RA and/or an interleukin-6 (IL-6) inhibitor for any purposes.
* Patient who has previously received more than 1 biologic agents approved for the treatment of RA.
* Patient who has allergies to any of the excipients of study drug or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The usability of AI as assessed by patients rating using POST-Self-Injection Assessment Questionnaire (SIAQ) at Week 2. | Week 2
  The POST-SIAQ module is a 27-item questionnaire that assesses feelings about injections, self-image, self-confidence, pain and skin reactions, ease of use and satisfaction with self-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Klimiuk Piotr, MD, PhD, Principal Investigator — INTER CLINIC Piotr Adrian Klimiuk

REFERENCES:
- [Derived] Burmester G, Klimiuk PA, Trefler J, Jaworski J, Kim S, Bae Y, Jeon D, Lee H, Jang J, Hwang C, Lee H, Smolen JS. Usability, efficacy, and safety of candidate tocilizumab biosimilar CT-P47 self-administration via auto-injector and pre-filled syringe in patients with rheumatoid arthritis: a single-arm, open-label, phase 3 study. Expert Rev Clin Immunol. 2025 Apr;21(4):521-529. doi: 10.1080/1744666X.2025.2451215. Epub 2025 Jan 15. PMID 39803727